CLINICAL TRIAL: NCT06449196
Title: An Experimental Medicine Vaccine Trial of Mosaic HIV-1 Envelope Trimer Immunogens Administered to People Living with HIV PLWH) in Africa, Randomized for Assessment of Fractional Doses
Brief Title: Mosaic HIV-1 Envelope Trimer Immunogens Administered to People Living with HIV (PLWH) in Africa
Acronym: C112
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Polymun Scientific GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IAVI C112
Record Dates: First submitted 2024-05-14; First posted 2024-06-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: HIV
Keywords: People Living with HIV (PLWH)
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bolus Dosing (Experimental): HIV Env Mosaic immunogens MOS1SIP, MOS2SIP, M3SIP8 and Monophosphoryl lipid A liposomes (MPLA-5) adjuvant (IM) administered via bolus dosing
  Interventions: Drug: Investigational product HIV Env Mosaic immunogens MOS1SIP, MOS2SIP, M3SIP8 and Monophosphoryl lipid A liposomes (MPLA-5) adjuvant (IM)
- Fractionated Dosing (Experimental): HIV Env Mosaic immunogens MOS1SIP, MOS2SIP, M3SIP8 and Monophosphoryl lipid A liposomes (MPLA-5) adjuvant (IM) administered via fractionated dosing
  Interventions: Drug: : Investigational product HIV Env Mosaic immunogens MOS1SIP, MOS2SIP, M3SIP8 and Monophosphoryl lipid A liposomes (MPLA-5) adjuvant (IM)

INTERVENTIONS:
Drug: Investigational product HIV Env Mosaic immunogens MOS1SIP, MOS2SIP, M3SIP8 and Monophosphoryl lipid A liposomes (MPLA-5) adjuvant (IM) — HIV Env Mosaic immunogens MOS1SIP, MOS2SIP, M3SIP8 and Monophosphoryl lipid A liposomes (MPLA-5) adjuvant (IM) administered via bolus dosing.
  Arms: Bolus Dosing
Drug: : Investigational product HIV Env Mosaic immunogens MOS1SIP, MOS2SIP, M3SIP8 and Monophosphoryl lipid A liposomes (MPLA-5) adjuvant (IM) — HIV Env Mosaic immunogens MOS1SIP, MOS2SIP, M3SIP8 and Monophosphoryl lipid A liposomes (MPLA-5) adjuvant (IM) administered via fractionated dosing
  Arms: Fractionated Dosing

SUMMARY:
An Experimental Medicine Vaccine Trial of Mosaic HIV-1 Envelope Trimer Immunogens Administered to People Living with HIV (PLWH) in Africa, Randomized for Assessment of Fractional Doses.

DETAILED DESCRIPTION:
The study will enroll people living with HIV, 18-50 years of age on a stable antiretroviral therapy regimen; principal exclusion criteria include history of AIDS-defining illness, significant acute or chronic medical condition other than HIV infection, and clinically significant laboratory abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV-1 infection (HIV Ab+ or HIV RNA+) by documentation in the medical records or in-clinic HIV testing;
2. CD4 ≥ 300 cells/µl;
3. Currently on ART, and documentation of continuous combination ART (cART) treatment with suppression of plasma HIV-1 viral load < 50 copies / ml for greater than 6 months, measured on at least 2 independent occasions, and with a viral load < 50 copies / ml at time of screening (within 42 days prior to IP administration). cART is defined as a regimen including ≥ 2 compounds, e.g., 2 nucleoside reverse transcriptase inhibitors plus either non nucleoside reverse transcriptase inhibitor or protease inhibitor or integrase inhibitor.
4. Having serum neutralization breadth of at least 20% using a 12-virus global panel at screening.
5. At least 18 years of age on the day of screening and has not reached his or her 51st birthday on the day of signing the Informed Consent Document.
6. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
7. In the opinion of the Principal Investigator or designee and based on Assessment of Informed Consent Understanding results, has understood the information provided and potential impact and/or risks linked to administration of the investigational product; written informed consent will be obtained from the participant before any study-related procedures are performed.
8. All sexually active female participants capable of becoming pregnant must commit to use an effective method of contraception for 4 months following IP administration, including:

   1. Condoms (male or female) with or without spermicide
   2. Diaphragm or cervical cap with spermicide
   3. Intrauterine device, or contraceptive implant
   4. Hormonal contraception
   5. Successful vasectomy in the male partner (considered successful if a woman reports that a male partner has [1] documentation of azoospermia by microscopy (< 1 year ago), or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post-vasectomy)
   6. Not be of reproductive potential, such as having undergone hysterectomy, bilateral oophorectomy, or tubal ligation, postmenopausal (>45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone [FSH] level >40 IU/L); surgically sterile: no additional contraception required.
9. Women, who are not sexually active at screening, must agree to utilize an effective method of contraception if they become sexually active, as outlined above. Note: The Sponsor considers the above methods of contraception to be effective. More restrictive measures may be required by the site.
10. All female participants must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Procedures and must test negative prior to IP administration.

Exclusion Criteria:

1. Any clinically significant acute or chronic medical condition, other than HIV infection, that is considered progressive or in the opinion of the investigator makes the participant unsuitable for participation in the study.
2. History of AIDS-defining illness or CD4 < 200 cells/µl.
3. If female, pregnant, lactating or planning a pregnancy during the period of screening through completion of the study.
4. In the past 6 months a history of alcohol or substance use, judged by the Investigator to potentially interfere with participant study compliance.
5. Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions). Note: A participant who states that he or she has easy bruising or bleeding but does not have a formal diagnosis and has intramuscular injections and blood draws without any adverse experience, is eligible.
6. History of a splenectomy.
7. Receipt of live attenuated vaccine within the previous 60 days or planned receipt within 60 days after administration of IP; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days of administration of the IP (exception is live attenuated influenza vaccine within 14 days).
8. Receipt of blood transfusion or blood-derived products within the previous 3 months.
9. Participation in another clinical trial of an investigational product currently, within the previous 3 months or expected participation during this study.
10. Prior receipt of an investigational HIV vaccine candidate, monoclonal antibody, or polyclonal immunoglobulin (note: receipt of placebo in a previous HIV vaccine or monoclonal antibody trial will not exclude a participant from participation if documentation is available and the Medical Monitor gives approval.
11. History of severe local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulties, angioedema);
12. Psychiatric condition that compromises safety of the participant and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
13. If, in the opinion of the Principal Investigator, it is not in the best interest of the participant to participate in the trial.
14. Seizure disorder: a participant who has had a seizure in the last 3 years is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years.)
15. Infectious disease: chronic hepatitis B infection (HbsAg), current hepatitis C infection (HCV Ab positive and HCV RNA positive) or treatment for hepatitis C infection in the past year, or active syphilis (RPR confirmed by TPHA).
16. A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy;
17. Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic, antiviral, or antifungal therapy within 30 days prior to enrolment.
18. Any of the following abnormal laboratory parameters listed below:

    Haematology
    * Haemoglobin <10.5 g/dL in females; haemoglobin <11.0 g/dL in males
    * Absolute Neutrophil Count (ANC): ≤1000/mm3
    * Absolute Lymphocyte Count (ALC): < 650/mm3
    * Platelets: < 125,000 mm3 or ≥ 550,000/mm3 Chemistry
    * Sodium ≤135 mEq/L or ≥ 146 mEq/L
    * Potassium ≤3.4 mEq/L or ≥ 5.6 mEq/L
    * Creatinine ≥1.1 x ULN
    * AST ≥1.25 x ULN
    * ALT ≥1.25 x ULN
    * Total bilirubin ≥1.25 x ULN
    * Alkaline phosphatase ≥1.25 x ULN
    * Albumin ≤ 3.0 g/dL or ≤ 30 g/L Urinalysis

    Clinically significant abnormal dipstick confirmed by microscopy:
    * Protein = 1+ or more
    * Blood = 1+ or more (not due to menses)
19. Any clinically relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease, other than HIV; use of systemic corticosteroids, immunosuppressive, anticancer, or other medications considered significant by the investigator within the previous 6 months.

The following exceptions are permitted and will not exclude study participation:

use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least 6 weeks prior to enrolment in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
To evaluate incidence of reactogenicity events, adverse events and serious adverse events (Safety and Tolerability). | 15 months
  Proportion of volunteers with moderate or greater reactogenicity events from initial administration through 7 days following completion of each dose of the investigational product.
  Proportion of volunteers with moderate or greater vaccine-related unsolicited adverse events (AEs), including safety laboratory (biochemical, hematological) parameters, from initial administration through 28 days following completion of each dose of the investigational product.
  Proportion of volunteers with vaccine-related serious adverse events (SAEs) throughout the study period.

SECONDARY OUTCOMES:
Immunogenicity | 15 months
  Proportion of volunteers with improvement in neutralizing activity, based on breadth and potency, prior to and after immunization with the Env Mosaic immunogens.
  Difference in neutralization breadth and potency with fractionated dosing compared to bolus doses of the Env Mosaic immunogens.
  Proportion, magnitude, and epitope-specificity of serum IgG binding responses to the Mosaic Env trimers after immunization with the Env Mosaic immunogens compared to baseline.

OTHER OUTCOMES:
Exploratory | 15 months
  Proportion of volunteers with improved breadth and potency of serum antibody neutralization against a tier 2 cross-clade global 12 virus panel of heterologous HIV-1 Env pseudotyped virus strains.
  Frequencies and phenotype of Env-specific plasmablast, germinal centre and memory B cells in peripheral blood mononuclear cells (PBMCs) and lymph node aspirates before and after immunization with Mosaic Env immunogens.

IPD SHARING:
Plan to Share IPD: Yes
This will be done with the clinical trial team, collaborators and funding agencies. Also, as information becomes available, this will be shared with the site and study participants. Results dissemination plans will be developed and implemented as the study progresses.
Supporting Information: Study Protocol
Time Frame: Information will be shared as soon as results are publicly available for the investigational product being used in similar studies conducted in other regions. The existing results and data upon which the C112 study is based is yet to be made fully publicly available.
Access Criteria: Access to data will be determined by the study team, partners and funding agencies.